CLINICAL TRIAL: NCT03970291
Title: Impact of Nociceptive-Level (NOL) Intraoperative Guided Fentanyl Analgesia Versus Standard Clinical Care (SCC) for Elective Major Abdominal Surgery
Brief Title: Impact of NOL Intraoperative Guided Fentanyl Analgesia vs SCC for Elective Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medasense Biometrics Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLI-01-1-08
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-07

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nociceptive-Level (NOL) (Experimental): Analgesic component of anesthesia (fentanyl) will be guided using NOL
  Interventions: Device: PMD-200
- Standard Clinical Care (SCC) (No Intervention): Standard Clinical Care guided fentanyl administration

INTERVENTIONS:
Device: PMD-200 — The PMD-200 system is comprised of a console and designated finger probe with 4 sensors. The Sensors are Photoplethysmography (PPG) Galvanic Skin Response (GSR), Accelerometer (ACC) and Thermistor (TMP)
  Arms: Nociceptive-Level (NOL)

SUMMARY:
Recently, a newly developed index, the Nociceptive Level (NOL) index, was validated and showed superiority over heart rate and blood pressure for recognition and grading of intense and mild nociceptive stimuli during surgery under general anesthesia.

We hypothesize that compared with standard management, NOL-guided anesthesia will lead to reduced postoperative pain scores, and during anesthesia, to increased hemodynamic stability.

DETAILED DESCRIPTION:
Uncontrolled postoperative pain may result in significant clinical, psychological, and socioeconomics consequences. Not only does inadequate pain management following surgery result in increased morbidity and mortality but it also may delay recovery, result in unanticipated readmissions, decrease patient satisfaction, and lead to chronic persistent postsurgical pain. Pain is multifactorial in nature and understanding both the complexity of pain and its side effects is imperative to achieve a successful surgical outcome.

Nociception/analgesia are currently assessed by monitoring changes in heart rate (HR), blood pressure (BP), and other indirect parameters which are not sensitive or specific to nociception. As a result, the patient may be given insufficient analgesia which can promote postoperative pain, or excessive analgesia which can result in overdosing and related complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old.
2. ASA I-III
3. Elective major laparoscopic abdominal surgical, urologic or gynecologic procedures under general anesthesia.
4. Patient able to provide informed consent

Exclusion Criteria:

1. Use of any type of anesthesia other than general anesthesia (neuraxial, epidural analgesia or local regional anesthesia, e.g. transversus abdominal plane block)
2. Patients with rhythm other than sinus cardiac rhythm, implanted pacemakers, α2-adrenergic agonists and β1-adrenergic antagonists
3. Pregnancy/lactation
4. Central nervous system disorder (neurologic/head trauma/uncontrolled epileptic seizures)
5. Abuse of alcohol or illicit drugs within the last 6 months
6. Chronic pain conditions - pain in 1 or more anatomic regions that persists or recurs for longer than 3 months and is associated with significant emotional distress or significant functional disability.
7. Opioid tolerant - if for at least 1 week the patient has been receiving oral morphine 60 mg/day; transdermal fentanyl 25 mcg/hour; oral hydromorphone 8 mg/day; oral oxymorphone 25 mg/day; or an equianalgesic dose of any other opioid
8. Chronic use of psychoactive drugs within 90 days prior to surgery
9. Allergy or intolerance to any of the study drugs
10. History of severe cardiac arrhythmias within the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Pain score | Through study completion, about 8 months
  Change in pain score in the PACU using the visual analog scale (VAS)

SECONDARY OUTCOMES:
Inadequate analgesia/anesthesia events | Through study completion, about 8 months
  Change in frequency of Inadequate analgesia/anesthesia events*
Total intraoperative fentanyl | Through study completion, about 8 months
  Change in total intraoperative fentanyl consumption (in mcg).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Rivka Leah Fuica, MD, Principal Investigator — Shaare Zedek
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuica R, Krochek C, Weissbrod R, Greenman D, Freundlich A, Gozal Y. Reduced postoperative pain in patients receiving nociception monitor guided analgesia during elective major abdominal surgery: a randomized, controlled trial. J Clin Monit Comput. 2023 Apr;37(2):481-491. doi: 10.1007/s10877-022-00906-1. Epub 2022 Aug 17. PMID 35976578